CLINICAL TRIAL: NCT03393247
Title: The Therapy Effect of Azathioprine Initial or 14 Weeks After Combined With Infliximab on Crohn Disease：a Randomized, Open Label, Single-center Cohort Study
Brief Title: The Therapy Effect of Azathioprine Initial or 14 Weeks After Combined With Infliximab on CD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSLY-XHNK-03
Record Dates: First submitted 2017-07-08; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-07

CONDITIONS: Crohn Disease
Keywords: infliximab; azathioprine
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- infliximab and azathioprine at week 0 (Active Comparator): infliximab and azathioprine combination at week 0
  Interventions: Drug: infliximab and azathioprine combination at week 0
- infliximab and azathioprine at week 14 (Active Comparator): infliximab and azathioprine combination at week 14
  Interventions: Drug: infliximab and azathioprine combination at week 14

INTERVENTIONS:
Drug: infliximab and azathioprine combination at week 0 — All enrolled CD patients will schedule on IF X (week 0, 2, 6 and then every 8 weeks at 5mg/kg).Experimental group will receive azathioprine at week 0.
  Arms: infliximab and azathioprine at week 0
Drug: infliximab and azathioprine combination at week 14 — All enrolled CD patients will schedule on IF X (week 0, 2, 6 and then every 8 weeks at 5mg/kg).Control group will receive azathioprine at week 14.
  Arms: infliximab and azathioprine at week 14

SUMMARY:
This study aim to identify the therapeutic effect of azathioprine during infliximab(IFX) treatment in Crohn's disease (CD).Half of patients will receive azathioprine and infliximab combination therapy at the same time. The other half patients will be given infliximab therapy first and then receive azathioprine 14 weeks later.

DETAILED DESCRIPTION:
Anti-tumor necrosis factor agents were widely used for many years and were proved to be most reliable drugs in Crohn's disease (CD). About one-third of the patients would develop a secondary lost of response after initiating IFX therapy in one year follow-up. Immunosuppressor was thought to be a useful agent to reduce loss of response rate of infliximab.But It remain unclear when should us add immunosuppressor during infliximab therapy.This study aim to find the most valuable timepoint to initiate combination therapy to maximize therapeutic effect and minimize the adverse effect.

ELIGIBILITY:
Inclusion Criteria:

- CD patients need infliximab and azathioprine combination therapy

Exclusion Criteria:

- patients had lost response to infliximab or azathioprine previously patients intolerable to infliximab or azathioprine patients need to use 5-Aminosalicylates(5-ASA) patients had participated to other clinical study in two months

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
loss of response(LOR) rate at one year | one year
  LOR was defined as recurrence or worsening of symptoms after achieving remission or response that required IFX dose intensification, addition of concomitant therapy, or discontinuation of IFX.

SECONDARY OUTCOMES:
Simple Endoscopic Score for Crohn's Disease(SES-CD) at one year | one year
  Patients will undergo colonscopy at one year after infliximab therapy and SES-CD which is a useful ool in evaluating endoscopic activities will be evaluated by colonoscopists.
Mucosal healing（MH）status at one year | one year
  Patients will undergo colonscopy at one year after infliximab therapy and mucosal healing（MH）means no ulcer in terminal ileum and colorectum.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Gao, doctor, Study Chair — the 6th affiliated hospital of Sun Yat-sen university
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided